CLINICAL TRIAL: NCT04206553
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Dupilumab in Adult Patients With Bullous Pemphigoid
Brief Title: A Study to Evaluate the Efficacy and Safety of Dupilumab in Adult Patients With Bullous Pemphigoid
Acronym: LIBERTY-BP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-BP-1902; 2019-003520-20 (EudraCT Number); 2024-510745-34-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — dupilumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dupilumab (Experimental)
  Interventions: Drug: dupilumab; Drug: Oral corticosteroids (OCS)
- Matching placebo (Experimental)
  Interventions: Drug: Matching Placebo; Drug: Oral corticosteroids (OCS)

INTERVENTIONS:
Drug: dupilumab — Loading dose administered subcutaneous (SC), followed by SC once every 2 weeks (Q2W) dosing.
  Other Names: Dupixent®; REGN668; SAR231893
  Arms: dupilumab
Drug: Matching Placebo — Matching dupilumab without active substance
  Arms: Matching placebo
Drug: Oral corticosteroids (OCS) — Prednisone or prednisolone per standard of care to obtain control of disease activity.

SUMMARY:
The main purpose of this study is to investigate whether dupilumab is effective and safe for the treatment of bullous pemphigoid. Dupilumab is a type of drug called a "monoclonal antibody". An antibody is a special kind of protein that the immune (defense) system normally makes to fight bacteria and viruses. Bullous pemphigoid is an autoimmune subepidermal blistering disease, predominately affecting the elderly (typical onset after age 60).

The study is looking at several other research questions, including:

* Side effects that may be experienced by people taking dupilumab
* How dupilumab works in the body and affects the body
* How dupilumab affects quality of life
* How much dupilumab is present in the blood
* To see if dupilumab works to wean the patient off oral corticosteroids

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must have characteristic clinical features of bullous pemphigoid (BP) (eg, urticarial or eczematous or erythematous plaques, bullae, pruritus) at the screening and baseline visits.
* Study participants are required to have a confirmed diagnosis of BP based on histopathology, immunopathology, and serology at the baseline visit, as defined in the protocol.
* Bullous Pemphigoid Disease Area Index (BPDAI) activity score ≥24 at baseline and screening visits.
* Baseline peak pruritus NRS score for maximum itch intensity ≥4
* Karnofsky performance status score ≥50% at the screening visit.

Key Exclusion Criteria:

* Forms of pemphigoid other than classic BP (eg, Brunsting-Perry cicatricial pemphigoid, anti-p200 pemphigoid, epidermolysis bullosa acquisita, or BP with concomitant pemphigus vulgaris)
* Patients who are receiving treatments known to cause or exacerbate BP (eg, angiotensin converting enzyme inhibitors, penicillamine, furosemide, phenacetin, dipeptidyl peptidase 4 inhibitor) who have not been on a stable dose of these medications for at least 4 weeks prior to the screening visit
* Have ever received treatment with an IL-4 or IL-13 antagonist such as dupilumab, tralokinumab, or lebrikizumab.
* Treatment with systemic corticosteroids within 7 days before the baseline visit
* Treatment with topical corticosteroids of medium potency or higher, topical calcineurin inhibitor, or topical crisaborole within 7 days before the baseline visit
* Treatment with non-steroidal immunosuppressive/immunomodulating drug(s) (eg, mycophenolate mofetil, azathioprine, or methotrexate) within 4 weeks before the baseline visit.
* Treatment with BP-directed biologics as follows:
* Any cell-depleting agents including but not limited to rituximab: within 12 months before the baseline visit, or until lymphocyte and CD 19+ lymphocyte count returns to normal, whichever is longer
* Other biologics (such as IL-5 inhibitors benralizumab or mepolizumab): within 5 half-lives (if known) or 16 weeks prior to the baseline visit, whichever is longer
* Intravenous immunoglobulin within 16 weeks prior to the baseline visit

NOTE: Other Protocol Defined Inclusion/Exclusion Criteria Apply

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving sustained remission | Week 36

SECONDARY OUTCOMES:
Total cumulative dose of oral corticosteroids (OCS) | Baseline to week 36
Percent change in weekly average of daily peak pruritus numerical rating score (NRS) | Baseline to week 36
  Individual NRS used to rate the intensity of pruritus using an 11-point scale (0 to 10) in which 0 indicates no itch while 10 indicates worst itch possible.
Proportion of patients with improvement (reduction) of weekly average of daily peak pruritus NRS ≥4 | Baseline to week 36
Percent change in Bullous Pemphigoid Disease Area Index Activity Score (BPDAI) activity score | Baseline to week 36
  BPDAI activity score is the arithmetic sum of 3 subcomponents: cutaneous blisters/erosions, cutaneous urticaria/erythema, and mucosal blisters/erosions. Scores can range from 0 to 360 for BPDAI total activity (maximum 240 for total skin activity and 120 for mucosal activity), with higher scores indicating greater disease activity.
Time to first use of rescue medication | Up to week 36

OTHER OUTCOMES:
Duration of complete remission while not requiring OCS | Baseline to week 36
Proportion of patients who do not achieve control of disease activity, who relapse after achieving control of disease activity, or do not achieve complete remission | Baseline to week 36
  Note: Control of disease activity is defined when new lesions cease to form and existing lesions begin to heal.
Proportion of patients who achieve a reduction in BPDAI activity score of at least 50%, 75%, and 90% | Baseline to week 36
Change in autoimmune bullous disease quality of life (ABQOL) | Baseline to week 36
  ABQOL questionnaire consists of 17 items, which encompass physical burden of the disease, psychiatric effects, and effects on daily life functioning. Each question ranges from 0 to 3 points, with higher scores indicating poorer quality of life. The maximum ABQOL score is 51.
Change in percent body surface area (BSA) of BP involvement | Baseline to week 36
Change in BP180 autoantibody (IgG) titers | Baseline to week 36
Change in BP230 autoantibody (IgG) titers | Baseline to week 36
Proportion of patients with sustained remission | Week 52
Total cumulative dose of OCS | Baseline to week 52
Duration of complete remission while not requiring OCS | Up to week 52
Proportion of patients who do not achieve control of disease activity, who relapse after achieving control of disease activity, or do not achieve complete remission | Up to week 52
Percent change in weekly average of daily peak pruritus NRS | Baseline to week 52
Proportion of patients with improvement (reduction) of weekly average of daily peak pruritus NRS ≥4 | Baseline to week 52
Percent change in BPDAI activity score | Baseline to week 52
Proportion of patients who achieve a reduction in BPDAI activity score of at least 50%, 75% and 90% | Baseline to week 52
Change in ABQOL | Baseline to week 52
Change in percent BSA of BP involvement | Baseline to week 52
Change in BP180 autoantibody (IgG) titers | Baseline to week 52
Change in BP230 autoantibody (IgG) titers | Baseline to week 52
Proportion of patients in complete remission and off OCS | Week 16
Percent change in BPDAI activity score | Baseline to week 16
Proportion of patients who achieve a reduction in BPDAI activity score of at least 50%, 75%, and 90% | Baseline to week 16
Percent change in weekly average of daily peak pruritus NRS | Baseline to week 16
Proportion of patients with improvement (reduction) of weekly average of daily peak pruritus NRS ≥4 | Baseline to week 16
Incidence of treatment-emergent adverse events (TEAEs) | Baseline to week 64
Incidence of treatment-emergent serious adverse events (SAEs) | Baseline to week 64
Incidence of adverse events of special interest (AESIs) | Baseline to week 64
Concentrations of functional dupilumab in serum | Baseline to week 64
Incidence of treatment-emergent anti-drug antibody (ADA) responses and titer | Baseline to week 64

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (53):
- United States (15):
  - Regeneron study Site, Birmingham, Alabama
  - Regeneron Study Site, Scottsdale, Arizona
  - Regeneron Study Site, Redwood City, California
  - Regeneron Study Site, Farmington, Connecticut
  - Regeneron Study Site, Miami, Florida
  - Regeneron study Site, Orlando, Florida
  - Regeneron Study Site, Iowa City, Iowa
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron study Site, Ann Arbor, Michigan
  - Regeneron Study Site, Chapel Hill, North Carolina
  - Regeneron Study Site, Portland, Oregon
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron study Site, Providence, Rhode Island
  - Regeneron Study Site, Murray, Utah
  - Regeneron study Site, Charlottesville, Virginia
- Australia (2):
  - Regeneron Study Site, Kogarah, New South Wales
  - Regeneron Study Site, Box Hill, Victoria
- France (6):
  - Regeneron Study Site, Bobigny
  - Regeneron Study Site, Bordeaux
  - Regeneron Study Site, Lille
  - Regeneron Study Site, Nice
  - Regeneron Study Site, Paris
  - Regeneron Study Site, Rouen
- Germany (12):
  - Regeneron Study Site, Münster, North Rhine-Westphal
  - Regeneron Study Site, Mainz, Rhineland-Palatinate
  - Regeneron Study Site 2, Dresden, Saxony
  - Regeneron Study Site, Lübeck, Schleswig-Holstein
  - Regeneron Study Site, Berlin
  - Regeneron Study Site, Buxtehude
  - Regeneron Study Site, Erlangen
  - Regeneron Study Site, Freiburg im Breisgau
  - Regeneron Study site', Magdeburg
  - Regeneron Study site, Marburg
  - Regeneron Study Site, Munich
  - Regeneron Study Site, Stuttgart
- Israel (3):
  - Regeneron study Site, Afula
  - Regeneron study Site, Petah Tikva
  - Regeneron study Site, Tel Aviv
- Japan (6):
  - Regeneron Study site, Kurume, Hukuoka
  - Regeneron Study Site, Hirosaki
  - Regeneron Study Site, Ichinomiya
  - Regeneron Study Site, Osaka
  - Regeneron Study Site, Sapporo
  - Regeneron Study Site, Tokyo
- Poland (3):
  - Regeneron Study Site, Krakow, Lesser Poland Voivodeship
  - Regeneron Study site', Ossy
  - Regeneron Study site', Wroclaw
- Spain (4):
  - Regeneron Study Site, Badalona, Barcelona
  - Regeneron Study Site, Madrid
  - Regeneron study Site, Madrid
  - Regeneron study Site, Pamplona
- Taiwan (2):
  - Regeneron study Site, Taipei, Zhongzheng District
  - Regeneron study Site, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Murrell DF, Joly P, Werth VP, Ujiie H, Worm M, Mangold AR, Avetisova E, Maloney J, Laws E, Mortensen E, Dubost-Brama A, Shabbir A. Study Design of a Phase 2/3 Randomized Controlled Trial of Dupilumab in Adults with Bullous Pemphigoid: LIBERTY-BP ADEPT. Adv Ther. 2024 Jul;41(7):2991-3002. doi: 10.1007/s12325-024-02810-3. Epub 2024 Mar 5. PMID 38443648